CLINICAL TRIAL: NCT06777862
Title: Investigation of Factors Affecting Quality of Life in Chronic Non-Specific Neck Pain
Brief Title: Chronic Non-Specific Neck Pain and Quality of Life
Status: Enrolling by invitation | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mensure Aslan, Physical Therapist, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-M.ASLAN-001
Record Dates: First submitted 2025-01-06; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Neck Pain; Quality of Life
Keywords: chronic neck pain; quality of life; depression; proprioception; muscle strength
MeSH Terms: conditions — Neck Pain; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The factors affecting the quality of life in individuals with chronic non-specific neck pain are not fully known in the studies conducted to date. The aim of this study was to examine the factors affecting the quality of life of individuals with chronic non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

No history of radicular pain, trauma or surgery in the cervical region,

* Between the ages of 18-65,
* Having neck pain for at least 6 months,
* Not having received any treatment for neck pain in the last year
* Volunteers with chronic non-specific neck pain

Exclusion Criteria:

* Those with any systemic disease
* Those with cervical pathology
* Previous surgery in the neck region
* Those with neuromuscular disease
* Those with rheumatology disease
* Infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of this study consists of individuals who applied to the Kırşehir Ahi Evran University Physical Medicine and Rehabilitation Polyclinic in Kırşehir province with complaints of neck pain and were diagnosed with chronic non-specific neck pain by specialist physicians.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-03 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
Pain Level | 6 weeks
  Visual Analog Scale (VAS) will be used to assess the severity of the patient's neck pain. The participant is asked to mark the severity of the pain on a 10-centimeter line (0=no pain, 10=very much pain)

SECONDARY OUTCOMES:
RANGE OF MOTION | 6 weeks
  Clinical goniometer will be used to measure the flexion, extension, lateral flexion and rotation range of motion of the cervical spine.
MUSCLE STRENGTH | 6 weeks
  In order to obtain objective data, maximal isometric muscle strength of the cervical region muscles will be measured with a Lafayette brand portable dynamometer. During the measurements, participants are asked to generate maximum force against the portable dynamometer device throughout the test (3-5 seconds).
Cervical Region Proprioception Sense | 6 weeks
  Joint position sense will be evaluated in four directions: left rotation, right rotation, extension and flexion with the Cervical Joint Position Sense Test. A total of ten measurements will be made, the first four for trial purposes. The average of the last six measurements will be taken for each direction.
Depression symptoms | 6 weeks
  Beck Depression Inventory (BDI) will be used to assess depression symptoms. The scale consists of 21 items, each of which is scored from 0 to 3. Higher scores indicate the severity of depression (1-10 points = normal, 11-16 points = moderate mood disturbance, 17-20 points = clinical depression, 21-30 points = moderate depression, 31-40 points = severe depression, 41-63 points = severe depression).
Quality of Life Level | 6 weeks
  The participants' quality of life will be assessed with the Short Form Health Survey -36 Quality of Life Scale. The scale consists of 36 statements and has 8 subheadings (physical function, pain, mental status, physical role limitation, emotional role limitation, vitality, social function and general perception of health). As the total score increases, the quality of life also increases. Scores for these scales are standardized into values ranging from 0 to 100 with 50 representing average health.
Sleep Quality | 6 weeks
  The participants' sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI). The scale consists of seven components (subjective sleep quality, time it takes to fall asleep, sleep duration, sleep disorders, use of medication for sleep, habitual efficiency of sleep and daily life dysfunction). Each component is valued between 0-5 points. The total score is 0-21 points (<5 points = good sleep quality, >5 points disturbed sleep quality).
Neck Disability Level | 6 weeks
  Neck Disability Questionnaire will be used to evaluate disability due to neck pain. The questionnaire consists of 10 questions. The questionnaire evaluates the intensity of pain in the neck region, difficulty in personal care and work, headache, pain level while reading, lifting performance, driving, difficulty level in sleeping and leisure activities. Each question is evaluated with 0-5 points and increasing score is associated with increasing disability. A high total score indicates that the individual's neck disability rate increases. (0-20 points = minimal disability, 21-40 points = moderate disability, 41-60 points = severe disability, 61-80 points = disability, 81-100 points = bedridden

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No